CLINICAL TRIAL: NCT07312695
Title: A Community Trial of Holly™ for Pediatric Populations in Naturalistic Settings
Brief Title: Holly™ Community Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Ontario Brain Institute (Other)
Responsible Party: Principal Investigator, Azadeh Kushki, Senior Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: eREB#0348
Record Dates: First submitted 2025-11-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Behavioural Responses and Emotional Reactivity
Keywords: wearable; emotion regulation; neurodevelopment disorder; anxiety
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- holly device trial (Experimental): Families try out holly™ at home, where the children will be given a study smartwatch with the holly™ app on it and asked to wear it for three weeks. Parents will get alerts and information about their child's emotional level on a study smartphone. Parents can use this information to help their child manage feelings as they happen. Parents can also use holly™ to review their child's emotion level history from the past day or days of use.
  Interventions: Device: holly device trial

INTERVENTIONS:
Device: holly device trial — Children will be given a study smartwatch with the holly™ app on it and asked to wear it for three weeks. Parents will get alerts and information about their child's emotional level on a study smartphone. Parents can use this information to help their child manage feelings as they happen. Parents can also use holly™ to review their child's emotion level history from the past day or days of use. Using holly, caregivers and children (where appropriate) will be provide with visualizations of arousal levels throughout the day and can be used to support children's emotional wellbeing.

SUMMARY:
This community study is a mixed effectiveness-implementation trial of holly™ for delivering information about arousal levels in paediatric populations. This study will evaluate the community implementation of holly™ and gather preliminary data on its impact on quality of life. holly™ is not meant to drive clinical decisions (diagnosis, monitoring, or intervention); instead, it is an informational tool to provide caregivers and children (where appropriate) with visualizations of arousal levels throughout the day and support children's emotional wellbeing.

For this study, the goal is to have families try out holly™ at home. The main objectives are:

1. To evaluate the implementation of holly™ in community settings. Specifically, A (primary)) To evaluate the usability of holly™ in community settings; and B) To evaluate the acceptability and adoption of holly™ in community settings.
2. To examine facilitators and barriers to real world implementation of holly™.

Exploratory Objective 1: To examine change (pre/post using holly™) in quality of life and mechanisms that may contribute to changes in quality of life (e.g., irritability, sleep, emotion regulation, anxiety, co-occurring symptoms).

Exploratory Objective 2: To gather preliminary data to explore associations between holly™ measurements and phenotypic and neurobiological characteristics to inform future trials and use cases.

holly™ is a patented and clinically validated algorithm for detecting emotional levels. Children will be given a study smartwatch with the holly™ application on it and asked to wear it for three weeks. Parents will get alerts and information about their child's emotional level on a study smartphone. Parents can use this information to help their child manage feelings as they happen. Parents can also use holly™ to review their child's emotion level history from the past day or days of use. Before and after using holly™, parents and children will be asked to fill out some questionnaires online. When families are finished with their three-week trial, they will be given a pre-paid shipping label to return the study devices to us.

ELIGIBILITY:
Inclusion Criteria:

* Strong emotional responses, such as outbursts, shutdowns, and/or meltdowns as reported by parents

Exclusion Criteria:

* Use of beta blockers

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Usability - System Usability Scale (SUS) | Post-intervention (up to 1 year after completion of the device trial period)
  To evaluate the usability of holly™ in community settings, the investigators will employ a summative evaluation approach through questionnaires. The primary measure will be the System Usability Scale (SUS), a 10-item parent questionnaire generating a score from 0-100 where higher is better. The criteria for success is an average score of 74 or higher on the SUS across the participants as per normative data for the SUS. Caregivers complete the measure following device usage.
Usability - Post-Study System Usability Questionnaire (PSSUQ) | Post-intervention (up to 1 year after completion of the device trial period)
  The Post-Study System Usability Questionnaire (PSSUQ) is a 16-item questionnaire that probes overall usability, system usefulness, information quality, and interface quality with acceptable estimated reliabilities of 0.83 to 0.96. Caregivers complete the measure following device usage.
  PSSUQ follows a 7-point Likert Scale (+ NA option). The overall result is calculated by averaging the scores from the 7 points of the scale. It has three sub-scales: system usefulness, information quality, and interface quality. The overall score can range from 1-7. The lower the score, the better the performance and satisfaction.
Usability - Custom Usability Questionnaire | Post-intervention (up to 1 year after completion of the device trial period)
  Children will complete a custom usability questionnaire assessing likeability and comfort of the smartwatch. The measure uses a visual Likert-type scale consisting of 3 items scored from 1 (lowest) to 3 (highest), with higher scores indicating better usability outcomes.
Acceptability and Adoption - Custom Parent Questionnaire | Post-intervention (up to 1 year after completion of the device trial period)
  The Custom Parent Questionnaire will measure users' intention to use holly™ after completion of the study, and extent to which holly™ was integrated in the users' lives, measured as the number of settings where holly™ is used during the trial (home, school, community). Caregivers complete the questionnaire following device usage.
Acceptability and Adoption - Client Satisfaction Questionnaire (CSQ-8) | Post-intervention (up to 1 year after completion of the device trial period)
  Acceptance, operationalized as the users' degree of satisfaction with holly™ and quantified using the Client Satisfaction Questionnaire (CSQ-8), an 8-item measure with high coefficients of internal consistency reliability (Cronbach's alpha of 0.80 or greater) and adequate validity. The instrument will be modified to include a description of the holly™ "service". Total scores range from 8 to 32, with the higher number indicating greater satisfaction. Caregivers complete the measure following device usage.
Acceptability and Adoption - Adapted version of the Barriers to Treatment Participation Scale | Post-intervention (up to 1 year after completion of the device trial period)
  To measure appropriateness, defined as the perceived fit, relevance, and compatibility of holly™ within the users' context, the investigators will be using an adapted version of the Barriers to Treatment Participation Scale, which demonstrates good psychometric properties regarding reliability and structure (internal consistency Cronbach's alpha of 0.85 or greater) and is reasonably valid. Caregivers complete this 32-item questionnaire rating of how much they agree with statements about their expectancies of barriers to treatment participation for their child, using a 5-point Likert scale (1=totally disagree, 5= totally agree). The total score ranges from 32 - 160, with higher score indicating greater barriers (i.e., worse outcome).
Acceptability and Adoption - Usage logs | During intervention (3-week device trial).
  The investigators will measure the number of hours holly™ is worn during the three-week trial, and rate of change in usage from week 1 to week 3. This information will be recorded by hollyTM.

OTHER OUTCOMES:
Relevance to Clinical Outcomes (Effectiveness) - Aberrant Behaviour Checklist (ABC-2) | Baseline and post-intervention (up to 1 year after completion of the device trial period).
  This measure will assess changes in irritability from pre- to post-device usage using the Aberrant Behaviour Checklist (ABC-2). Participants complete the ABC-2 at enrollment (baseline) and again immediately after completing the device trial period. The ABC-2 is a validated caregiver-reported measure of problem behaviours in individuals with neurodevelopmental conditions. It uses a 4-point Likert scale to score aberrant behaviors, where 0 is "not a problem" and 3 is "severe problem". Scores are summed for each of the five subscales: irritability, social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech. The possible total is between 0-174 and a higher score indicates worse outcome.
Relevance to Clinical Outcomes (Effectiveness) - Children's Sleep Habit Questionnaire (CSHQ) | Baseline and post-intervention (up to 1 year after completion of the device trial period). For POND study participants, baseline CSHQ collected at enrollment, or existing POND CSHQ collected within the last two years.
  This measure will assess changes in sleep habits from pre- to post-device usage using the Children's Sleep Habit Questionnaire (CSHQ). Caregivers complete the CSHQ at enrollment (baseline) and again immediately after the device trial period. The CSHQ is a validated caregiver-reported measure of sleep behaviors in children, capturing domains such as bedtime resistance, sleep duration, night wakings, and daytime sleepiness. The total possible score ranges from 33-99, with higher score indicating worse outcome.
  For participants who previously completed the CSHQ as part of the POND study at Holland Bloorview, existing data will be retrieved with participant consent (signed Release of Information) if collected within the last two years; otherwise, the measure will be repeated.
Relevance to Clinical Outcomes (Effectiveness) - Emotion Dysregulation Inventory (EDI) | Baseline and post-intervention (up to 1 year after completion of the device trial period).
  This measure will assess changes in emotion regulation abilities from pre- to post-device usage using the Emotion Dysregulation Inventory (EDI). Caregivers complete the EDI at enrollment (baseline) and again immediately after the device trial period. The EDI is a validated caregiver-reported measure designed to capture reactivity and dysregulation in children with neurodevelopmental conditions. The EDI uses a 5-point scale for items of problem severity over the past 7 days, where 0 = not at all a problem and 4 = very severe problem. It is scored on two subscales: Reactivity (intense emotional reactions) and Dysphoria (sadness, low motivation). Raw scores from the 24-item Reactivity scale (min = 0 and max = 96) or 6-item Dysphoria scale (min = 0 and max = 24) can be converted to t-scores for comparison against different population norms, such as a general youth sample or a clinical sample for individuals with autism. Higher scores indicate worse outcomes.
Relevance to Clinical Outcomes (Effectiveness) - Pediatric Quality of Life Inventory (PedsQL) | Baseline and post-intervention (up to 1 year after completion of the device trial period).
  The Pediatric Quality of Life Inventory (PedsQL) will be used to evaluate changes in health-related quality of life from baseline to post-device usage. Caregivers will complete the age-appropriate version of the PedsQL (Young Child 5-7 years, Child 8-12 years, or Teen 13+ years) at enrollment and again immediately after the device trial period.
  Each PedsQL form uses a 5-point response scale (0-4) that is converted to a 0-100 scale, with higher scores indicating better outcomes (i.e., better health-related quality of life). Subscale and total scores will be calculated according to standardized PedsQL scoring procedures.
Relevance to Clinical Outcomes (Effectiveness) - Parent Rated Anxiety Scale in ASD (PRAS-ASD) | Baseline, and post-intervention (up to 1 year after completion of the device trial period).
  This measure will assess changes in anxiety levels from pre- to post-device usage using the Parent Rated Anxiety Scale in ASD (PRAS-ASD). Caregivers complete the PRAS-ASD at enrollment (baseline) and again immediately after the device trial period. The PRAS-ASD is a validated caregiver-reported measure designed to capture anxiety symptoms specifically in autistic children. It is a 25-item, parent-report questionnaire where item is rated on a 0-3 scale, with a total raw score ranging from 0 to 75. Higher score indicates worse outcome.
Exploration of associations with phenotypic and neuroimaging profiles - Neuroimaging data | At study completion, using previously collected POND neuroimaging data when available.
  The investigators will examine associations between phenotypic measures and neuroimaging profiles using existing structural MRI, diffusion tensor imaging, and resting-state data from the Province of Ontario Neurodevelopmental Disorders (POND) Network. With participant consent (signed Release of Information), neuroimaging data previously collected by the POND study will be retrieved when available.
Arousal Variables: Mean Heart Rate During Device Usage | During the intervention (3-week device trial)
  This measure will summarize average heart rate recorded by the holly device during usage period. Heart rate data will be used to examine physiological arousal patterns over the trial period, along with other arousal variables, and to characterize changes across the trial period and to explore associations with phenotypic and neuroimaging profiles.
Arousal VariablesHeart Rate Variability During Device Usage | During intervention (3-week device trial)
  This measure will summarize heart rate variability (HRV) obtained from the holly device during usage periods. HRV will be analyzed as an indicator of autonomic arousal, along with other arousal variables, and used to characterize changes across the trial period and to explore associations with phenotypic and neuroimaging profiles.
Arousal Variable: Number of Arousal Events During Device Usage | During intervention (3-week device trial)
  This measure will record the count of physiological arousal events detected by the holly device during usage. Event counts will be evaluated over the trial period along with other arousal variables to characterize changes across the trial period and to explore associations with phenotypic and neuroimaging profiles.
Arousal Variables: Mean Acceleration During Device Usage | During intervention (3-week device trial)
  This measure will summarize the average acceleration recorded by the holly device to summarize physiological arousal during device usage. Mean acceleration values, along with other arousal variables, will be used to characterize changes across the trial period and to explore associations with phenotypic and neuroimaging profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Kushki, PhD., Principal Investigator — Hollanf Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No